CLINICAL TRIAL: NCT00426582
Title: A Phase Ib, Multicenter, Open-label, Dose-finding Study of Patupilone Administered Intravenously Every 3 Weeks in Combination With Carboplatin AUC 6 in Adult Patients With Advanced Solid Tumors
Brief Title: Combination Trial of Patupilone and Carboplatin in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2105
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2011-03

CONDITIONS: Advanced Solid Tumors
Keywords: Cancer; maximum tolerated dose; dose-limiting toxicity; patupilone; carboplatin; pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — epothilone B

ARMS (2):
- Patupilone only (Experimental): Cycle 1 patupilone alone Cycle 2 and onward patupilone and carboplatin
  Interventions: Drug: Patupilone
- Carboplatin alone (Active Comparator): Cycle 1 Carboplatin alone Cycle 2 and onward patuilone and carboplatin
  Interventions: Drug: Patupilone

INTERVENTIONS:
Drug: Patupilone

SUMMARY:
This study will evaluate the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of patupilone combined with carboplatin in adult patients with advanced solid tumors who progressed despite standard therapy or for whom no standard therapy exists or who might benefit from treatment with carboplatin

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed advanced solid tumors who have progressed despite standard therapy, or for whom no standard therapy exists, or who might benefit from treatment with carboplatin
* A minimum of 4 weeks since the last treatment with chemotherapy
* WHO Performance Status 0 (able to carry out all normal activity without restriction) or 1 (restricted in physically strenuous activity but ambulatory and able to carry out work)
* Age ≥ 18
* Adequate hematological parameters
* No major impairment of renal or hepatic function
* Written informed consent obtained

Exclusion criteria:

* Major surgery less than 4 weeks prior to study entry and/or not fully recovered from surgery
* Chemotherapy or investigational compound less than 4 weeks prior to study entry, or planned while participating in the study
* Prior administration of an epothilone
* Hypersensitivity to carboplatin. Patients resistant to carboplatin are not recommended to enter the trial
* Radiotherapy (RT) less than 4 weeks prior to study entry (except for palliative therapy of distant metastases), or planned RT while participating in the study
* Diarrhea within 7 days prior to start of treatment. Unresolved bowel obstruction
* Peripheral neuropathy > Grade 1 (mild)
* Symptomatic brain metastases
* Colostomy

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-08; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of patupilone in combination with carboplatin (AUC 6) | Every 3 weeks

SECONDARY OUTCOMES:
Safety of patupilone combined with carboplatin assessed by adverse events, serious adverse events, laboratory values and physical examinations | Every 6 weeks
Overall response rate (complete and partial response; CR + PR) according to RECIST (response evaluation criteria in solid tumors) | Every 6 weeks
Time to progression (TTP), duration of overall response, duration of stable disease and time to overall response | Every 6 weeks
Pharmacokinetic profile of patupilone combined with carboplatin | First 6 weeks (cycle 1 & 2 only)
Relationship between pharmacokinetics and clinical outcome | Every 6 weeks during cycle 1 & cycle 2

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (5):
- United States (5):
  - Norwalk Hospital, Norwalk, Connecticut
  - Associates in Oncology, Rockville, Maryland
  - Wertz Clinical Cancer Center (Wayne State University), Detroit, Michigan
  - Siteman Cancer Center (Washington University School of Medicine), St Louis, Missouri
  - Cancer Research and Treatment Center (University of New Mexico), Albuquerque, New Mexico

REFERENCES:
- See also: Results can be found for CEPO906A2105 on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5244